CLINICAL TRIAL: NCT00145015
Title: Fish Consumption and Gastro-Intestinal Health With Special Emphasis on Reduction of Risk of Colon Cancer and Inflammatory Bowel Disease
Brief Title: FishGastro Study: Fish Consumption and Gastro-Intestinal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Wageningen University (Other); University of Jena (Other); University of East Anglia (Other); European Commission (Other); Food Standards Agency, United Kingdom (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IFR02/2004
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Colorectal Cancer; Ulcerative Colitis; Polyps
Keywords: Intervention; Adults; Colorectal cancer; Nutrition; Fish; n-3 fatty acids; Apoptosis; Ulcerative colitis; Polyps; Gastro-intestinal tract
MeSH Terms: conditions — Colorectal Neoplasms; Colitis, Ulcerative; Polyps | interventions — CVD protocol

INTERVENTIONS:
Behavioral: Increased dietary intake of salmon or cod

SUMMARY:
The purpose of the study is to determine whether increasing the dietary intake of n-3 fatty acids by the consumption of oil-rich fish reduces the risk of developing colorectal cancer.

DETAILED DESCRIPTION:
Epidemiological evidence from several countries supports a protective effect of fish consumption on cancer risk and gastrointestinal cancers in particular. Further evidence to support the idea that fish consumption is protective in relation to cancers of the GI tract is now emerging from the European Investigation into Cancer and Nutrition (EPIC).

The FISHGASTRO project is headed by the Institute of Food Research and includes groups from the University of East Anglia, the University of Wageningen, Netherlands and the University of Jena, Germany. The project focuses on assessing the impact of fish consumption on a range of markers of gastrointestinal health associated with ulcerative colitis or colon cancer and on looking at bio-accessibility of a range of nutrients from fish. We aim to recruit a total of 270 patients with gastrointestinal problems in the UK and Netherlands and take biopsy and blood samples before and after asking them to eat two extra portions of fish per week. One group will receive oil rich fish such as salmon while another will be asked to eat white fish. Changes in cell proliferation, apoptosis, inflammatory markers, gene expression and plasma levels of n-3 fatty acids will be compared to a control group only given standard nutritional advice.

ELIGIBILITY:
Inclusion Criteria:

Ulcerative Colitis Patient Group (Group 1):

* Aged 18 - 80
* Male or female
* Diagnosed with ulcerative colitis
* Attending gastroenterology clinic for routine colonoscopy check-up
* Willing to increase dietary intake of fish for six months
* Willing to undergo a flexible sigmoidoscopy examination

Polyps/Resection Group (Group 2):

* Aged 18 - 80
* Male or female
* A history of polyps in the colon
* Attending gastroenterology clinic for routine colonoscopy check-up
* Willing to increase dietary intake of fish for six months
* Willing to undergo a flexible sigmoidoscopy examination

Control Group (Group 3):

* Aged 18 - 80
* Male or female
* Booked for a colonoscopy examination for the investigation of iron deficiency anaemia of unknown cause (no evidence of macroscopic disease found during examination)
* Willing to increase dietary intake of fish for six months
* Willing to undergo a flexible sigmoidoscopy examination

Exclusion Criteria:

Ulcerative Colitis Patient Group (Group 1) and Polyps/Resection Group (Group 2):

* Allergic to fish
* Receiving anticoagulant therapy
* Diabetics
* Pregnant or breast-feeding
* Organ transplant recipients receiving immunosuppression therapy
* Prosthetic heart valve
* Allergic to pethidine
* Previous diagnosis of bacterial endocarditis

Control Group (Group 3):

Same as Groups 1 and 2 plus:

* Received a diagnosis of colorectal cancer following initial investigative colonoscopy (volunteer will be withdrawn from the study when diagnosed as requiring treatment)
* Received a diagnosis of coeliac disease following initial investigative colonoscopy (volunteer will be withdrawn from the study when diagnosed as requiring a modified diet)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2004-12; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Apoptosis in colonic biopsy samples

SECONDARY OUTCOMES:
Cell proliferation
lymphocyte infiltration
circulating inflammatory markers (cytokines and prostaglandins)
tissue inflammatory markers (cytokines and prostaglandins)
faecal water cytotoxicity and genotoxicity
gene transcription

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Lund, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (2):
- University of Wageningen, Wageningen, Netherlands
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Pot GK, Geelen A, Majsak-Newman G, Harvey LJ, Nagengast FM, Witteman BJ, van de Meeberg PC, Hart AR, Schaafsma G, Lund EK, Rijkers GT, Kampman E. Increased consumption of fatty and lean fish reduces serum C-reactive protein concentrations but not inflammation markers in feces and in colonic biopsies. J Nutr. 2010 Feb;140(2):371-6. doi: 10.3945/jn.109.113472. Epub 2009 Dec 23. PMID 20032491
- [Derived] Pot GK, Majsak-Newman G, Geelen A, Harvey LJ, Nagengast FM, Witteman BJ, van de Meeberg PC, Timmer R, Tan A, Wahab PJ, Hart AR, Williams MP, Przybylska-Phillips K, Dainty JR, Schaafsma G, Kampman E, Lund EK; FISHGASTRO Study Group. Fish consumption and markers of colorectal cancer risk: a multicenter randomized controlled trial. Am J Clin Nutr. 2009 Aug;90(2):354-61. doi: 10.3945/ajcn.2009.27630. Epub 2009 Jun 24. PMID 19553301